CLINICAL TRIAL: NCT03856671
Title: Prophylatic Effect of Preoperative Antibiotics With Mechanical Bowel Preparation Compare With Simple Mechanical Bowel Preparation Before Laparoscopic Colorectal Surgery: a Randomized Controlled Trial
Brief Title: Prophylatic Effect Preoperative Antibiotics With Mechanical Bowel Preparation in SSIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OAMBP-01
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Surgical Site Infection; Postoperative Complications; Bowel Preparation; Oral Antibiotics; Colorectal Cancer
Keywords: Surgical Site Infection; oral antibiotics; mechanical bowel preparation; laparoscopic surgery
MeSH Terms: conditions — Surgical Wound Infection; Postoperative Complications; Colorectal Neoplasms | interventions — Neomycin; Metronidazole

STUDY DESIGN:
Masking Description: No masking is to conducted in the current study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral antibiotics+mechanical bowel preparation (Experimental): Liquid diet and polyethylene glycol with 2L water was administrated orally 1 day before surgery. A combination of neomycin 1g and metronidazole 0.2g every 6 hours was also administrated. Enteroclysis was conduted for patients on surgical morning.
  Interventions: Drug: Neomycin,metronidazole
- simple mechanical bowel preparation (No Intervention): Only liquid diet and polyethylene glycol with 2L water was administrated orally 1 day before surgery. Enteroclysis was conduted for patients on surgical morning.

INTERVENTIONS:
Drug: Neomycin,metronidazole — Orally intake neomycin 1g and metronidazole 0.2g four times before surgery
  Arms: oral antibiotics+mechanical bowel preparation

SUMMARY:
Surgical site infection (SSI) is a major postoperative complication after abdominal surgery especially in colorectal field, which significantly increases length of stay (LOS), readmission incidence and expense. Therefore, identification of the effective method to reduce SSI incidence is critically important. Combination of oral antibiotics and mechanical bowel preparation was reported with lower SSIs and LOS in some retrospecitve data analysis, however a prospective randmized controlled trial was absent. Herein, the current randomized controlled trial comparing MBP+OA with MBP alone in postoperative complications in order to guide clinical practise was conducted.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is a major postoperative complication after abdominal surgery especially in colorectal field, which significantly increases length of stay (LOS), readmission incidence and expense. Therefore, identification of the effective method to reduce SSI incidence is critically important. Colonic bacterial flora is the major cause of SSIs after elective colorectal procedures. For more than century, preoperative mechanical bowel preparation (MBP) has been utilized as it could theoretically decrease bacterial load within the surgical field, thus reduce risk of SSIs. Later afterwards with widely application of antibiotics, combination of oral antibiotics (OA) and MBP was conducted by surgeons to further decrease rates of SSIs. But SSIs still occurs despite of forehead mentioned methods, the best bowel preparation mode remains controversial. Since 2005, several RCTs and meta-analysises demonstrated MBP alone was not associated with reduced SSIs compared with no bowel preparation, while postoperative ileus, anastomotic leakage and other complications incidence increased paradoxically. Nevertheless, function of preoperative oral antibiotics remains debated. Recently, combination of oral antibiotics and MBP has been evaluated in several retrospective studies and demonstrated a significant decrease in the rate of SSIs. However, bias existence in these trials may affect result as information was exacted from national database without detailed matching. Herein, current randomized controlled trial comparing MBP+OA with MBP alone in postoperative complications in order to guide clinical practise was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old，
* Undergoing laparoscopic colorectal surgery due to malignancy.

Exclusion Criteria:

* No elective surgery
* Intra-abdominal infection
* Combination of other infectious surgery such as appendectomy, cholecystomy
* Sever comobidity such as uncontrolled hypertention and diabetes mellitus
* Peritoneal implantation and matastasis
* Radiotherapy history.
* Colorectal surgery due to benign lesions
* Allergic to antibiotics or PEG
* Preoperative dermatosis may interfere wound healing
* Long time application of corticosteroid
* Autoimmune disease may affect wound healing
* Patients refuse to enroll

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Surgical site infection incidence | 30 days after surgery
  Include the superficial, deep and organ space infection.

SECONDARY OUTCOMES:
Antibiotics associated complications | 30 days after surgery
  Allergy, antibiotics associated diarrhea
Length of hospital stay after surgery | 30 days after surgery
  Length of hospital stay
Bowel recovery time | 7 days after surgery
  Time interval from surgery to flatus and defecation
Other posteroperative complications | 30 days after surgery
  Ilues, DVT, anastomotic fistula, hemorrhage, pulmonary infection

CONTACTS AND LOCATIONS:
Overall Officials: Hongbo Wei, Ph.D, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-Sen university, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lei P, Jia G, Yang X, Ruan Y, Wei B, Chen T. Region-specific protection effect of preoperative oral antibiotics combined with mechanical bowel preparation before laparoscopic colorectal resection: a prospective randomized controlled trial. Int J Surg. 2023 Oct 1;109(10):3042-3051. doi: 10.1097/JS9.0000000000000569. PMID 37702427
- [Derived] Willis MA, Toews I, Soltau SL, Kalff JC, Meerpohl JJ, Vilz TO. Preoperative combined mechanical and oral antibiotic bowel preparation for preventing complications in elective colorectal surgery. Cochrane Database Syst Rev. 2023 Feb 7;2(2):CD014909. doi: 10.1002/14651858.CD014909.pub2. PMID 36748942